CLINICAL TRIAL: NCT03334227
Title: High Flow Nasal Cannula Therapy as an Adjuvant in the Treatment of Severe Sepsis. A Multicenter Parallel-group Randomized Clinical Trial
Brief Title: High Flow Nasal Cannula in Severe Sepsis
Acronym: OPTISEPSIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Rafael Fernandez, Director. Critical Care Department, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI17/54
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Severe Sepsis
Keywords: High-Flow Nasal Cannula; Severe Sepsis; qSOFA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Patients with severe sepsis will be randomized to recieve conventional oxygenotherapy if needed or high flow nasal cannula.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Flow nasal cannula (HFNC) (Experimental): Treatment with HFNC will be adjusted for SpO2 >92%, even with FiO2 of 0.21, if needed.
  The rationale for this HFNC dosage is that minute ventilation can be already reduced with 30 L/min, but functional residual capacity and oxygenation maximally improve at higher flow. On the contrary, flow >50 L/min is uncomfortable for many patients.
  In the case of clinical intolerance, flow will be reduced to 40, 30 or 20 L/min. Yet it is not tolerated, HFNC will be stopped and patients will receive conventional oxygen if required, but will be evaluated as in the HFNC group by intention to treat.
  Interventions: Device: High-Flow nasal cannula (HFNC)
- Conventional therapy (No Intervention): Patients assigned to the conventional treatment will receive the standard care given at hospital which consists of adding oxygen on nasal prongs or Venturi mask only if hypoxemia is suggested by SpO2 < 92% by pulse oximetry.
  Target for oxygenation in both arms is SpO2 between 92% and 95%. SpO2 >95% without oxygen supply is acceptable. On the contrary, SpO2 <92% may be acceptable when needed for medical reasons, mainly chronic hypercapnic patients.

INTERVENTIONS:
Device: High-Flow nasal cannula (HFNC) — The patient will receive HFNC adjusted for SatO2 > 92% and with, at least, 30 liters of total flow.
  Other Names: Conventional therapy
  Arms: High-Flow nasal cannula (HFNC)

SUMMARY:
Severe sepsis leads a high morbidity and mortality by causing organ damage at distance. The treatment relies on early antibiotic therapy and hemodynamic resuscitation. Hypothesis: high flow nasal cannula (HFNC) could reduce work of breathing and improve the outcome of patients with severe sepsis and peripheral perfusion. Objective: the aim of this study is to evaluate the efficacy of HFNC for improving sixty-day survival in patients with severe sepsis. Design: multicenter parallel-group randomized clinical trial. Method: 592 adult patients with a diagnosis of severe sepsis in the first 12 hours of admission in the Emergency Room will be randomly assigned to an experimental or control group. In the experimental group, HFNC will be administered until the resolution of sepsis or until required mechanical ventilation, either invasive or non-invasive. In the Control group, conventional oxygen will be administered, if required. Sixty-day survival will be the primary outcome. The study is powered to demonstrate an improvement in survival from 70% in control group up to 80% in the HFNC group. The secondary outcomes will be reducing the need for vital support (mechanical ventilation, dialysis, vasoactive drugs) and physiological (acidosis, clearance of lactate, SvO2 and SOFA). Statistical analysis: Kaplan-Meier curves and Cox proportional hazard models will be calculated for all-cause sixty-day survival. If the results are conclusive, they will have immediate application in medical practice.

DETAILED DESCRIPTION:
Severe sepsis is a syndrome associated with severe infections with a high morbidity and mortality. In its most severe form, septic shock still leads to an in-hospital mortality of up to 50%. The pathophysiology of severe sepsis / septic shock includes increased work of breathing to compensate for tissue hypoperfusion-induced metabolic acidosis. This exaggerated work of breathing requires increased consumption of oxygen by respiratory muscles, which calls for a greater percentage of the already insufficient cardiac output, which can aggravate tissue hypoperfusion.

In the last decade, high flow nasal cannula (HFNC) appeared as an alternative ventilatory support intermediate between conventional oxygen and mechanical ventilation. Among others (3-7), the investigators have also demonstrated their effectiveness in patients with respiratory failure of different etiologies (8-11). Patients treated with HFNC quickly show a reduction of respiratory rate and respiratory work, associated with an improvement of the functional residual capacity and gas exchange. The absence of significant side effects and low cost makes HFNC especially attractive as adjunctive medical treatment in severe sepsis.

Then, the hypothesis is that in patients with severe sepsis, high flow nasal cannula (HFNC) therapy could reduce work of breathing, which would allow a redistribution of cardiac output from the respiratory muscles to other organs, improving peripheral perfusion with minor injury of organs at distance, less multiorgan failure and improved survival. Therefore, the aim of this study is to evaluate the efficacy of HFNC for improving sixty-day survival in patients with severe sepsis. This study will also provide a detailed evaluation of the HFNC's effects on the need for vital support (mechanical ventilation, dialysis, vasoactive drugs) and physiological parameters (acidosis, clearance of lactate, SvO2 and SOFA).

DESIGN Prospective, multicenter, randomized, controlled trial in 592 patients with severe sepsis admitted into a network of 18 ICUs from university and community hospitals in Spain to define the role of high flow oxygen therapy, with one experimental arm that will receive high flow oxygen therapy and a control arm that will receive conventional oxygen therapy if required.

Patients who consent will be randomized in a 1:1 ratio to receive HFNC or conventional treatment, which consists of adding oxygen on nasal prongs or Venturi mask only if hypoxemia is detected as SpO2 < 92% by pulse oximetry.

STUDY ARMS

1. HFNC therapy (experimental group) Treatment with HFNC (Airvo2® Fisher & Paykel, and AquaNASE® Armstrong Medical) will begin with high flow (50 L/min), high temperature and humidity and oxygen concentration adjusted for SpO2 >92%, even with FiO2 of 0.21, if needed.

   The rationale for this HFNC dosage is that minute ventilation can be already reduced with 30 L/min, but functional residual capacity and oxygenation maximally improve at higher flow. On the contrary, flow >50 L/min is uncomfortable for many patients.

   In the case of clinical intolerance, flow will be reduced to 40, 30 or 20 L/min. Yet it is not tolerated, HFNC will be stopped and patients will receive conventional oxygen if required, but will be evaluated as in the HFNC group by intention to treat.

   In HFNC patients we propose an extra caution to avoid delaying a mechanical ventilation that would be beneficial. To do this, the ROX index (ROX = SpO2/FiO2/respiratory rate) will be calculated and if it is < 5, it is recommended to assess mechanical ventilatory support, either invasive or non-invasive.
2. Conventional therapy (control group) Patients assigned to the conventional treatment will receive the standard care given at hospital which consists of adding oxygen on nasal prongs or Venturi mask only if hypoxemia is suggested by SpO2 < 92% by pulse oximetry.

Target for oxygenation in both arms is SpO2 between 92% and 95%. SpO2 >95% without oxygen supply is acceptable. On the contrary, SpO2 <92% may be acceptable when needed for medical reasons, mainly chronic hypercapnic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 yr. with diagnostic criteria for severe sepsis, within 12 hours of admission in the Emergency Room, defined as hypotension after hemodynamic resuscitation, initial lactate > 4, or persistence of organ dysfunction (oliguria < 0.5 ml/kg/h, cyanosis, or altered consciousness).(qSOFA 1, 2 or 3)

Exclusion Criteria:

* Patients who require immediate ventilatory support both invasive and non-invasive, defined by severe hypoxemia (PaO2/FiO2 < 150), severe tachypnea (40 x') with signs of respiratory fatigue or low level of consciousness (Glasgow < 8).
* Patients with limitation of the therapeutic effort or orders of not CPR.
* Patients not susceptible to treatment with HFNC (facial trauma, tracheostomized, rejection of previous treatments with HFNC).
* Participation in other clinical trials that may affect survival.
* Home treatment with oxygen, CPAP or Non-invasive ventilation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Mortality | 60 day
  60-day survival after enrollment

SECONDARY OUTCOMES:
Mechanical ventilation support | up to 60-days
  Institution of mechanical ventilation (either invasive or noninvasive)
Dialysis support | up to 60-days
  Institution of dialysis
Vasoactive drugs tappering | up to 60-days
  Daily dose of vasoactive drugs until stopping
Sequential Organ Failure Assessment | up to 60-days
  Daily Sequential Organ Failure Assessment score. The organs scored are respiratory, cardiovascular, neurologic, hematologic, renal, and liver. Each organ is scored as 0 (best) to 4 (worse) and the total score is the sum of each component.
Acidosis improvement | up to 60-days
  Hours until the ph becomes normal
Central Venous Oxygen Saturation (SatVO2) | up to 60-days
  Hours until the SatVO2 < 65%
Lactate clearance | up to 60-days
  Hours until lactate < 3 mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, PhD, Principal Investigator — Fundacio Althaia
Locations (1):
- ICU. Fundacio Althaia, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Result] Viires N, Sillye G, Aubier M, Rassidakis A, Roussos C. Regional blood flow distribution in dog during induced hypotension and low cardiac output. Spontaneous breathing versus artificial ventilation. J Clin Invest. 1983 Sep;72(3):935-47. doi: 10.1172/JCI111065. PMID 6886012
- [Result] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Result] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Result] Stephan F, Barrucand B, Petit P, Rezaiguia-Delclaux S, Medard A, Delannoy B, Cosserant B, Flicoteaux G, Imbert A, Pilorge C, Berard L; BiPOP Study Group. High-Flow Nasal Oxygen vs Noninvasive Positive Airway Pressure in Hypoxemic Patients After Cardiothoracic Surgery: A Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2331-9. doi: 10.1001/jama.2015.5213. PMID 25980660
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Result] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Result] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Result] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461